CLINICAL TRIAL: NCT06621485
Title: Multi-institutional Development and Validation of an Individualized Online Calculator for Early Mortality Risk After Hepatectomy Among Patients With Hepatocellular Carcinoma
Brief Title: Calculator Predicts Early Mortality Post Hepatocellular Carcinoma Resection
Status: Completed | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Collaborators: Eastern Hepatobiliary Surgery Hospital of Shanghai (Unknown); The First Hospital of Jilin University (Other); Mengchao Hepatobiliary Hospital (Unknown); The Fourth Affiliated Hospital of Harbin Medical University (Other); Pu'er People's Hospital (Unknown); Liuyang People's Hospital (Unknown); Ziyang First People's Hospital (Unknown); Qianfoshan Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); Fuyang people's hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 24467-4-01
Record Dates: First submitted 2024-09-29; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: To Predict Early Post-hepatectomy Mortality for HCC
Keywords: Hepatocellular carcinoma; Hepatectomy; Survival; Morbidity; Futile surgery
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort: The training cohort was comprised of patients from 9 participating hospitals (First Hospital of Jilin University, Mengchao Hepatobiliary Hospital, the Fourth Hospital of Harbin, Pu'er People's Hospital, Liuyang People's Hospital, Ziyang First People's Hospital, First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, First Affiliated Hospital of Harbin Medical University, and Fuyang People's Hospital).
- Validation cohort: The validation cohort consisted of patients from the remaining two hospitals (Beijing Tsinghua Changgung Hospital and Eastern Hepatobiliary Surgery Hospital of Shanghai)

SUMMARY:
Using the multicenter data, we developed and validated an individualized online calculator to predict early mortality after liver resection for hepatocellular carcinoma. The user-friendly tool with 6 preoperative predictors demonstrated excellent accuracy. The freely available calculator may help identify high-risk patients and reduce futile liver resection for hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

Adults (age ≥18 years) who underwent curative-intent hepatectomy for newly diagnosed HCC.

HCC diagnosis was confirmed histopathologically.

Exclusion Criteria:

Patients undergoing emergency hepatectomy for tumor rupture, as well as individuals with recurrent HCC, and those with missing survival data or less than 90 days of follow-up were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The final analytic cohort was comprised of 4,966 HCC patients treated with hepatectomy with curative intent across 11 hospitals; 3,433 patients were in the 9-center training cohort and 1,533 in the 2-center external validation cohort.
Sampling Method: Non-Probability Sample
Enrollment: 4966 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
90-day death | The period starts from the day of the hepatectomy surgery and extends up to the 90th day post-surgery.
  90-day mortality after hepatectomy for HCC

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No